CLINICAL TRIAL: NCT00236145
Title: A Randomised, Open-label, Parallel-group Study to Evaluate the Efficacy and Safety of ACTIQ (Oral Transmucosal Fentanyl Citrate) Titrated According to 2 Regimens in Patients With Cancer and Breakthrough Pain
Brief Title: Evaluate the Efficacy and Safety of ACTIQ in Patients With Cancer and Breakthrough Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C8278A/302/ON/MN
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2005-10

CONDITIONS: Breakthrough Pain
Keywords: BTP; Break through pain; breakthrough pain
MeSH Terms: conditions — Breakthrough Pain | interventions — Fentanyl

INTERVENTIONS:
Drug: ACTIQ (Oral transmucosal fentanyl citrate)

SUMMARY:
The primary objective of the study is to determine whether a test titration regimen of ACTIQ treatment will reduce the number of inadequately managed episodes of breakthrough pain for an individual patient by attaining a successful dose of ACTIQ treatment more quickly. The successful ACTIQ dose provides a satisfactory combination of efficacy and tolerability after a single administration, as assessed by the patient.

ELIGIBILITY:
Inclusion Criteria: Patients are included in the study if all of the following criteria are met:

* the patient is at least 18 years old
* women must be surgically sterile, 2 years postmenopausal, or if of child-bearing potential, must use a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device)
* the patient experiences persistent pain associated with cancer or cancer treatment
* for at least 7 days before enrolment, the patient has taken either the equivalent of 60 to 1000 mg/day of oral morphine around-the-clock (ATC) or 25 to 300 micrograms/hr of transdermal fentanyl to treat persistent pain
* the patient regularly experiences between 1 and 4 episodes of cancer-related BTP per day while taking ATC opioid therapy
* the patient experiences at least partial relief of cancer related BTP by administering conventional opioid BTP medication at a dose approximately in the range of one-fifth to one-sixth the 24-hour sustained release dose
* the patient is capable of self-administering ACTIQ by sucking lozenge, producing sufficient saliva to dissolve the lozenge over 15 minutes, and swallowing the saliva
* a responsible adult caregiver is available to assist the patient in case of emergency if the patient will be taking ACTIQ at home
* the patient willingly provides informed consent to participate in this study

Exclusion Criteria: Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* the patient experiences uncontrolled or rapidly escalating pain, as determined by the investigator, such that ATC administration of pain medication might be expected to change between the first and last administrations of ACTIQ.
* the patient has known or suspected hypersensitivities and/or allergies to fentanyl
* the patient has a recent history or current evidence or abuse of alcohol or any other drug substance, licit or collection
* the patient has neurological or psychiatric disease sufficient, in the investigator's opinion, to compromise data collection
* the patient received strontium-89 therapy within 6o days prior to entering the study
* the patient received any other therapy (eg, radiotherapy) within a 1 week period prior to entering the study that, in the investigator's opinion, could alter pain or response to pain medication
* the patient has moderate to severe oral mucositis
* the patient is pregnant, nursing, or is of child-bearing potential or not taking adequate contraceptive measures
* the patient has previously been treated with ACTIQ
* the patient has participated in a trial of an unapproved drug in the previous 8 weeks
* the patient has been diagnosed with either severe respiratory depression or severe obstructive lung conditions
* the patient has used monoamine-oxidase inhibitors (MAOI's) within the 2-week period prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
to determine if ACTIQ treatment will reduce the number of inadequately managed episodes of breakthrough pain